CLINICAL TRIAL: NCT07379229
Title: Investigation of the Relationship Between Cognitive and Functional Status in Geriatric Patients With Hand-Forearm Injuries
Brief Title: The Cognitive-Functional Relationship in Geriatric Hand-Forearm Injuries
Status: Not yet recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, UMUT ERASLAN, Assistant Professor, Pamukkale University
Other Study IDs: E-60116787-020-808743
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Geriatric Population; Cognitive Ability; Functional Abilities; Hand Injuries
Keywords: geriatric population; hand Injuries; functional outcome; cognitive function
MeSH Terms: conditions — Hand Injuries | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Geriatric patients with hand-forearm injuries
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Injury severity will be assessed using the Modified Hand Injury Severity Score. At week 12 after the injury or surgery, cognitive status by Mini-Mental Test, upper extremity function by Upper Extremity Functional Index, pain intensity by Visual Analog Scale, and grip-pinch strength will be evaluated.

SUMMARY:
Considering the complex structure of hand-forearm injuries and the long rehabilitation process, it is important to investigate factors associated with recovery in geriatric individuals. Therefore, this study aimed to examine the relationship between cognitive status and functional outcomes in geriatric individuals with hand-forearm injuries.

ELIGIBILITY:
Inclusion Criteria:

* Being over 65 years of age
* Having sufficient communication skills and auditory-visual abilities to complete cognitive tests

Exclusion Criteria:

* Inability to perform functional tests due to active wounds, open fractures, or severe pain
* Inability to administer cognitive tests due to aphasia or severe hearing or visual impairment

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Volunteer geriatric individuals who were treated conservatively or surgically for hand and forearm injuries at the hand surgery clinic of a university hospital, and who were referred to the hand rehabilitation unit will be included.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Modified Hand Injury Severity Score | At baseline
  A scoring system that evaluates the severity of hand and forearm injuries based on integumentary, skeletal, motor, and neurovascular components. The total score is obtained by summing the scores of all components and is divided into four categories: minor (<20), moderate (21-50), severe (51-100), and major (>101) injury.
Standardized Mini-Mental Test | At 12th week after injury or surgery
  This test will be used to assess the cognitive levels of the participants. The test consists of five subdomains: orientation, registration, attention and calculation, recall, and language, and is scored out of a total of 30 points. The results are evaluated as follows; 27-30 points: within normal limits, 24-27 points: mild cognitive impairment, and below 24 points: severe cognitive impairment.
Upper Extremity Functional Index | At 12th week after the injury or surgery
  A 20-item scale used to assess upper extremity function and is scored using a 0-5 Likert-type rating, with a total score ranging from 0 to 80. Lower scores indicate that the individual has difficulty performing activities as a result of an upper extremity problem.
Grip-pinch strength | At 12th week after injury or surgery
  Grip strength will be measured using a Jamar hand dynamometer according to the procedure recommended by the American Society of Hand Therapists. Pinch strength will be measured using a Jamar pinch gauge in four positions: tip pinch, pulp pinch, lateral pinch, and tripod pinch. Results will be recorded in kilograms.
Perceived pain intensity | At 12th week after injury or surgery
  Perceived pain intensity will be assessed using the Visual Analog Scale. The evaluation will be performed on a 10-cm line ranging from "no pain" to "worst possible pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Carrillo CB, Barr C, George S. Cognitive Status and Outcomes of Older People in Orthopedic Rehabilitation? A Retrospective-Cohort Study. Geriatrics (Basel). 2020 Mar 2;5(1):14. doi: 10.3390/geriatrics5010014. PMID 32131454
- [Result] Kringstad O, Dahlin LB, Rosberg HE. Hand injuries in an older population - a retrospective cohort study from a single hand surgery centre. BMC Musculoskelet Disord. 2019 May 24;20(1):245. doi: 10.1186/s12891-019-2617-x. PMID 31122232